CLINICAL TRIAL: NCT07138183
Title: The Impact of Nurse Practitioner-Led Multidisciplinary Team Intervention on the Implementation of Guideline-Directed Medical Therapy and Clinical Outcomes in Adults With Multimorbidity: A Randomized Controlled Trial
Brief Title: The Impact of Nurse Practitioner-Led Multidisciplinary Team Intervention on the Implementation of Guideline-Directed Medical Therapy and Clinical Outcomes in Adults With Multimorbidity
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Clinical Trial Center, Principal Investigator, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202506113RINC
Record Dates: First submitted 2025-08-05; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Multimorbidity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NP-led MDT Intervention Group (Experimental): Participants receive care from a nurse practitioner-led multidisciplinary team providing individualized, guideline-based medication recommendations.
  Interventions: Behavioral: NP-led MDT
- Usual Care Group (Active Comparator): Participants receive usual inpatient care from the primary care team without additional NP-led MDT intervention.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: NP-led MDT — a nurse practitioner-led multidisciplinary team (MDT).
  Arms: NP-led MDT Intervention Group
Behavioral: Usual Care — Participants will receive usual inpatient care provided by the primary care team.
  Arms: Usual Care Group

SUMMARY:
The goal of this clinical trial is to evaluate whether a nurse practitioner-led multidisciplinary team (NP-led MDT) intervention can improve the use of guideline-directed medical therapy (GDMT) and short-term clinical outcomes in hospitalized adults with multimorbidity in a multidisciplinary medicine ward.

The main questions it aims to answer are:

Does NP-led MDT intervention increase the proportion of patients achieving GDMT at hospital discharge?

Does NP-led MDT intervention reduce 30-, 60-, and 90-day readmission, emergency department visits, and mortality?

Researchers will compare the NP-led MDT intervention group with the usual care group to see if the intervention improves GDMT implementation and clinical outcomes.

Participants will:

Be randomly assigned to NP-led MDT care or usual care.

Have their medications reviewed according to the latest guidelines (intervention group only).

Be followed for 90 days after discharge to collect outcomes through medical record review and telephone follow-up.

DETAILED DESCRIPTION:
This is a prospective, single-center, randomized controlled trial designed to evaluate whether a nurse practitioner-led multidisciplinary team (NP-led MDT) intervention can improve the implementation rate of guideline-directed medical therapy (GDMT) and short-term clinical outcomes in hospitalized adults with multimorbidity. Multimorbidity is defined as the coexistence of two or more chronic conditions, including heart failure, hypertension, diabetes mellitus, chronic kidney disease, ischemic heart disease, and chronic obstructive pulmonary disease. Suboptimal use of GDMT is common in this population, contributing to poor clinical outcomes.

Eligible patients admitted from the emergency department to the multidisciplinary medicine ward of a tertiary medical center will be screened within 72 hours of admission. Participants will be randomly assigned in a 1:1 ratio to either the NP-led MDT intervention group or the usual care group.

In the intervention group, the NP-led MDT-comprising a nurse practitioner, physicians, and clinical pharmacists-will review each patient's diagnoses, comorbidities, baseline medications, and relevant laboratory or imaging results. Based on the latest international guidelines, the team will formulate individualized GDMT recommendations, which will be communicated to the patient's primary inpatient care team. The NP will also provide patient and caregiver education on medication adherence, potential side effects, and follow-up requirements. All final prescribing decisions will be made by the primary physician.

In the usual care group, patients will receive standard inpatient management from their primary care team without additional structured NP-led MDT intervention.

The primary outcome is the GDMT implementation rate at hospital discharge, calculated as the number of GDMT drugs prescribed divided by the number indicated according to guidelines. Secondary outcomes include all-cause readmission, emergency department visits, and mortality at 30, 60, and 90 days post-discharge, as well as selected disease-specific clinical indicators when available (e.g., left ventricular ejection fraction, HbA1c, blood pressure, LDL-C, eGFR).

Follow-up will be conducted via medical record review and telephone contact. This trial aims to provide real-world evidence on whether an NP-led MDT approach can bridge the gap between guideline recommendations and actual prescribing practices, thereby improving both medication use and patient outcomes in multimorbid inpatients.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 years or older
2. Admitted to the multidisciplinary ward through the emergency department for inpatient care
3. Diagnosed with at least one of the following six chronic conditions and concurrently having one or more additional chronic diseases:

   * Congestive Heart Failure (CHF)
   * Diabetes Mellitus (DM)
   * Hypertension (HTN)
   * Dyslipidemia (DLP)
   * Atrial Fibrillation (AF)
   * Chronic Kidney Disease (CKD)

Exclusion Criteria:

1. End-of-life (EOL) patients: Refers to patients receiving palliative care or those assessed by the medical team as unlikely to survive to discharge during the current hospitalization.
2. Patients expected to be transferred to other departments: For example, patients anticipated to be transferred to oncology, intensive care unit (ICU), surgery, or other departments where full MDT intervention cannot be implemented.
3. Unwilling to participate.
4. Patients under the care of the study team physician on the day of hospitalization.
5. Patients known to be economically or educationally disadvantaged

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
GDMT Implementation Rate at Hospital Discharge | On the day of hospital discharge
  The proportion of guideline-directed medical therapy (GDMT) drugs prescribed at hospital discharge, calculated as the number of GDMT drug classes prescribed divided by the number of drug classes indicated.

CONTACTS AND LOCATIONS:
Overall Officials: Hsiao-Chen Chou Nurse Practitioner, Principal Investigator — National Taiwan University Hospital

IPD SHARING:
Plan to Share IPD: No
The individual participant data will not be shared due to patient privacy concerns and institutional policy restrictions. Only aggregated study results will be made publicly available.

REFERENCES:
- [Background] Spahillari A, Cohen LP, Lin C, Liu Y, Tringale A, Sheppard KE, Ko C, Khairnar R, Williamson KM, Wasfy JH, Scott NS, Paquette C, Greene SJ, Fonarow GC, Januzzi JL Jr. Efficacy, Safety and Mechanistic Impact of a Heart Failure Guideline-Directed Medical Therapy Clinic. JACC Heart Fail. 2025 Apr;13(4):554-568. doi: 10.1016/j.jchf.2024.08.017. Epub 2024 Oct 9. PMID 39387769
- [Background] AlHabeeb W, Alayoubi F, Hayajneh A, Ullah A, Elshaer F. A strategy to improve adherence to guideline-directed medical therapy (GDMT) and the role of the multidisciplinary team in a heart-failure programme. Cardiovasc J Afr. 2024 Jan-Apr 23;35(1):12-15. doi: 10.5830/CVJA-2022-067. Epub 2023 May 5. PMID 37171293
- [Background] Rao VU, Bhasin A, Vargas J Jr, Arun Kumar V. A multidisciplinary approach to heart failure care in the hospital: improving the patient journey. Hosp Pract (1995). 2022 Aug;50(3):170-182. doi: 10.1080/21548331.2022.2082776. Epub 2022 Jul 4. PMID 35658810
- [Background] Kidney Disease: Improving Global Outcomes (KDIGO) CKD Work Group. KDIGO 2024 Clinical Practice Guideline for the Evaluation and Management of Chronic Kidney Disease. Kidney Int. 2024 Apr;105(4S):S117-S314. doi: 10.1016/j.kint.2023.10.018. No abstract available. PMID 38490803
- [Background] Huang PH, Lu YW, Tsai YL, Wu YW, Li HY, Chang HY, Wu CH, Yang CY, Tarng DC, Huang CC, Ho LT, Lin CF, Chien SC, Wu YJ, Yeh HI, Pan WH, Li YH; expert committee for the Taiwan Lipid Guidelines for Primary Prevention. 2022 Taiwan lipid guidelines for primary prevention. J Formos Med Assoc. 2022 Dec;121(12):2393-2407. doi: 10.1016/j.jfma.2022.05.010. Epub 2022 Jun 14. PMID 35715290
- [Background] Wang TD, Chiang CE, Chao TH, Cheng HM, Wu YW, Wu YJ, Lin YH, Chen MY, Ueng KC, Chang WT, Lee YH, Wang YC, Chu PH, Chao TF, Kao HL, Hou CJ, Lin TH. 2022 Guidelines of the Taiwan Society of Cardiology and the Taiwan Hypertension Society for the Management of Hypertension. Acta Cardiol Sin. 2022 May;38(3):225-325. doi: 10.6515/ACS.202205_38(3).20220321A. PMID 35673334
- [Background] Joglar JA, Chung MK, Armbruster AL, Benjamin EJ, Chyou JY, Cronin EM, Deswal A, Eckhardt LL, Goldberger ZD, Gopinathannair R, Gorenek B, Hess PL, Hlatky M, Hogan G, Ibeh C, Indik JH, Kido K, Kusumoto F, Link MS, Linta KT, Marcus GM, McCarthy PM, Patel N, Patton KK, Perez MV, Piccini JP, Russo AM, Sanders P, Streur MM, Thomas KL, Times S, Tisdale JE, Valente AM, Van Wagoner DR; Peer Review Committee Members. 2023 ACC/AHA/ACCP/HRS Guideline for the Diagnosis and Management of Atrial Fibrillation: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. Circulation. 2024 Jan 2;149(1):e1-e156. doi: 10.1161/CIR.0000000000001193. Epub 2023 Nov 30. PMID 38033089
- [Background] Li YH, Wang CC, Hung CL, Wu YW, Hsu CH, Tsou YL, Wang CH, Wu CK, Lin PL, Chang HY, Sung SH, Chen ZW, Juang JJ, Wang TD, Chen WJ. 2024 Guidelines of the Taiwan Society of Cardiology for the Diagnosis and Treatment of Heart Failure with Preserved Ejection Fraction. Acta Cardiol Sin. 2024 Mar;40(2):148-171. doi: 10.6515/ACS.202403_40(2).20240206A. PMID 38532817